CLINICAL TRIAL: NCT06212843
Title: Effect of 8 Week Plyometric Training on Injury Prevention in Domestic Cricket Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 014241 aqsa safdar
Record Dates: First submitted 2023-11-25; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Injury Prevention
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Plyometric training) (Experimental)
  Interventions: Other: plyometric training
- Group B (Conventional) (Other)
  Interventions: Other: conventional exercises

INTERVENTIONS:
Other: plyometric training — The group will receive plyometric exercises in a controlled environment. Following Plyometrics would be performed.
  1. Plyo Pushup.
  2. Chest Pass.
  3. Overhead Throw.
  4. Squat jump.
  5. Plyo Step-up.
  6. Cone jumps.
  7. Med Ball drop.
  8. Kneeling Squat jump.
  9. Lateral jump over hurdle.
  10. Overhead throw.
  11. Under hand throws.
  12. Dynamic Rotational Chest pass.
  13. Overhead throw with step.
  Arms: Group A (Plyometric training)
Other: conventional exercises — The group will receive conventional exercises in a controlled environment. Following conventional exercises would be performed.
  1. Pushups.
  2. Situps.
  3. Lunges 4.500m running.
  5.Squats
  Arms: Group B (Conventional)

SUMMARY:
The study aims to find the effectiveness of plyometric training on injury prevention of domestic cricket players. Players will be taken from Chakwal and a well designed plyometric plan will be implied on them for 8 weeks. After that the results will be compared with the other group who did not get any plyometric training to see the effectiveness of the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* domestic cricket players between 18-25 years.
* actively engaged for more than 1 year

Exclusion Criteria:

* history of trauma/injury in last month

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Deep squat Test | 8 weeks
  The deep squat test typically involves a qualitative assessment rather than a numerical score. Trained evaluators observe the individual's form during the squat, looking for deviations such as heels lifting, knees collapsing, or torso leaning forward. A smooth, controlled movement with proper alignment is considered optimal. Interpretation involves identifying any biomechanical issues, muscle imbalances, or flexibility limitations based on observed deviations. This qualitative information guides fitness professionals, coaches, or healthcare providers in tailoring corrective exercises or interventions to address specific movement patterns or limitations identified during the deep squat test.
One legged squat | 8 weeks
  The one-legged squat, also known as the single-leg squat or pistol squat, is a functional movement exercise that challenges lower body strength, balance, and flexibility. In this exercise, an individual stands on one leg while lowering their body into a squat position and then returning to the starting position. Scoring typically involves assessing the ability to maintain balance, depth of the squat, and overall control during the movement. Interpretation focuses on identifying any asymmetries, weaknesses, or compensations in the lower body, helping tailor specific exercises or interventions to improve strength and stability in the individual's functional movement patterns.
Inline lunges | 8 weeks
  The inline lunge is a functional movement assessment used to evaluate lower body flexibility, balance, and symmetry. In this exercise, an individual steps forward into a lunge position along a straight line, assessing the ability to maintain proper alignment and stability. Scoring involves observing the quality of the lunge, noting any deviations or asymmetries in movement. Interpretation focuses on identifying potential issues in hip, knee, or ankle mobility, as well as muscle imbalances. The inline lunge is often employed in fitness and rehabilitation settings to tailor targeted exercises or interventions for improving lower body function and reducing the risk of injury.
active hip flexion test | 8 weeks
  The Active Hip Flexion Test is a functional movement assessment that evaluates the flexibility and mobility of the hip flexors. In this test, an individual lies on their back and actively lifts one leg straight up towards their chest while keeping the opposite leg flat on the surface. The angle of hip flexion is measured, and any limitations or discomfort are noted. Scoring involves assessing the range of motion, and interpretation focuses on identifying potential hip flexor tightness or restrictions. This test is commonly used in fitness, sports, and rehabilitation settings to inform targeted exercises or interventions aimed at improving hip flexor flexibility and function.
straight leg raise test | 8 weeks
  The Straight Leg Raise (SLR) Test is a clinical assessment used to evaluate the flexibility and tension of the hamstrings and the sciatic nerve. In this test, an individual lies on their back, and one leg is lifted upward while keeping the knee straight. The angle at which the leg can be raised before experiencing discomfort or tension is measured. Scoring involves noting the range of motion, and interpretation focuses on identifying potential issues such as hamstring tightness or sciatic nerve irritation.
Push-up | 8 weeks
  The push-up test is a fitness assessment that measures upper body strength and endurance. During the test, individuals perform as many push-ups as possible while maintaining proper form, including a straight body alignment. The number of completed push-ups is recorded, and interpretation varies based on age, gender, and fitness level norms.
Diagonal lift | 8 weeks
  The Diagonal Lift Test is a functional movement assessment that evaluates the coordination and stability of the core and lower body. In this test, an individual stands on one leg and lifts the opposite leg diagonally across the body. The goal is to perform the movement smoothly and with control. Scoring involves observing balance, fluidity, and any compensations or asymmetries. Interpretation focuses on identifying potential weaknesses, imbalances, or mobility restrictions in the core and lower extremities.
Seated rotation test | 8 weeks
  functional movement to help identify compensatory movement pattern and limitation
functional shoulder mobility | 8 weeks
  The Functional Shoulder Mobility Test is an assessment that evaluates the range of motion and flexibility in the shoulders, emphasizing their functional capacity. During the test, individuals perform various shoulder movements, such as reaching overhead, across the body, and behind the back. Scoring involves observing the range of motion, symmetry, and any discomfort or restrictions in the movements.

CONTACTS AND LOCATIONS:
Overall Officials: Aqsa safdar, DPT, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Riphah international university, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No